CLINICAL TRIAL: NCT03344315
Title: Xenogeneic Collagen Matrix or Palatal Connective Tissue Graft With a Coronally Advanced Flap for the Treatment of Miller Class III Gingival Recessions
Brief Title: Xenogeneic Collagen Matrix or Palatal Connective Tissue Graft With a Coronally Advanced Flap in Class III Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Elena Ruiz de Gopegui Palacios, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017_02
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Gingival Recession
Keywords: Gingival recession; Collagen matrix; Connective tissue graft; Coronally advanced flap; Root coverage; keratinized tissue; Periodontal disease
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Outcomes Assessor
Masking Description: Observer: Another periodoncist outside the intervention, would be in charge of recording the clinical parameters.
  Analyst: The statistician does not know which treatment corresponds to each variable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- autologous connective tissue graft (Active Comparator): Soft tissue harvesting from patient palate
  Interventions: Other: Active Comparator: autologous connective tissue graft
- collagen matrix (Experimental): Mucograft collagen matrix manufactured by Geistlich AG, Switzerland Device: Collagen matrix
  Interventions: Device: experimental: collagen matrix

INTERVENTIONS:
Device: experimental: collagen matrix — Mucograft collagen matrix combined with coronal advanced flap
  Arms: collagen matrix
Other: Active Comparator: autologous connective tissue graft — Soft tissue harvesting from patient palate with coronal advanced flap
  Arms: autologous connective tissue graft

SUMMARY:
The purpose of this multi-center study is to compare the effectiveness of Mucograft versus connective tissue graft in combination with coronal advanced flap for the treatment of Miller class III recessions The connective tissue graft in combination with coronal advanced flap is considered the gold standard for the treatment of gingival recession in terms of percentage of root coverage and complete root coverage. However connective tissue graft harvesting from the palatal mucosa is often associated with increased patient morbidity, prolonged surgical time and is limited supply. To overcome these inconvenients many efforts are made to develop new materials (healing modifiers, barrier membranes and grafts substitutes) Recently a new two-layer , xenogenic collagen matrix (Mucograft: Geistlich Pharma , Wolhusen Switzerland) has been proposed for regenerative therapy involving teeth and implants. The use of this porcine collagen matrix has obtained promising results for treatment of Miller class I and II recession defects (isolated and multiple recession defects) The mayority of root coverage studies in the literature treats Miller class I and II recession defects .Surgical treatment of class III recesión defects is more challenging due to loss of interproximal bone and soft tissues and complete root coverage may not be expected . But some recent studies demonstrate complete root coverage and high percentage of root coverage in class III recessions. Also a new classification system using the level of interproximal attachment level has been proposed to predict the final root coverage outcome.

So ,the soft tissue substitutes should be used also in Miller class III recession, and because of that fact, the investigators are conducting this study, to evaluate the effectiveness of Mucograft in Miller class III recessions compared with connective tissue graft.

DETAILED DESCRIPTION:
Given data reported by the study of Aroca in 2013 ,using the percentage of root coverage as a primary response variable the sample size was estimated in 20 patients. In addition, taking into account possible drop-outs, the investigators would increase the number of patients by 20%, finally recruiting 24 patients per group.

Randomization was performed by computer generated random codes Study locations will include two private centers in Spain. A single calibrated examiner, blind with respect to the treatment assignment, will perform all measurements at all center.

A biostatistician blind with respect to treatment assignment will perform the analysis.

Interventions and Duration The two intervention groups will consist of surgery with connective tissue graft (standard of care control) and surgery with the application of Mucograft Collagen Matrix (MCM, Test group). Experienced clinicians will deliver treatment consisting of root coverage surgery using coronally advanced flaps, the most utilized procedure for coverage of recessions. Surgery will be standardized and the same procedures/materials will be employed to ensure consistency.

Follow-up of individual patients will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years or older
* Patient with one or more recession defects are Miller Class III in incisives, canines and premolars. In at least two quadrants
* Patient shows sufficient plaque control (FMPS < 20%).
* Treated periodontal conditions
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent.

Exclusion Criteria:

* General contraindications for dental and/or surgical treatment are present.
* The patient is taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs).
* Untreated periodontal conditions
* Patients not willing to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years to 75 years
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage | Change from baseline at following surgery sixth and twelfth month respectively
  In each patient the mean of their gingival recessions at baseline (initial RECm)and at 6 (RECm 6months)and 12 months (RECm 12 months) will be calculated measuring at the mid buccal point of the involved teeth by the same blinded investigator using the same periodontal probe (PCP SE-11 Hu Friedly, Chicago, IL USA). With this measurements the percentage of root coverage will be calculated

SECONDARY OUTCOMES:
Percentage of recessions with Complete root coverage | Change from baseline at following surgery sixth and twelfth month respectively
  The number of recessions which after the treatment show complete root coverage (no recession) measured at the mid buccal point of the involved teeth at baseline and at 6 and 12 months .
Patient centred outcomes | after surgery up to 7 days and 1 year
  At suture removal both procedures will be evaluated by the patient for discomfort, duration and difficulty on a visual analogue scale (VAS) . At 12 months the aesthetic outcome obtained with both treatment modalities will be appreciated by the patient on a VAS scale.
Gingival Thickness | Change from baseline at following surgery and twelfth month respectively
  The thickness in millimeters measured 3mm apically from the free gingival margin at the mid buccal aspect of the tooth
Keratinized Tissue width | Change from baseline at following surgery sixth and twelfth month respectively
  Distance from the mucogingival junction to the gingival margin
Clinical Attachment Level | Change from baseline at following surgery sixth and twelfth month respectively
  The gain of clinical attachment level in milimetres, compared with baseline
Recession width | Change from baseline at following surgery sixth and twelfth month respectively
  Mesio-distal distance taken in the coronal area of the same, measured in millimeters.
Aesthetic results | 12 months
  The same blinded investigator will measured the aesthetic result by using the root coverage esthetic score system (RES)
Time of surgery | After surgery up to 7 days
  At surgery, the length of time of the full procedure will be evaluated (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Aguirre Zorzano, Principal Investigator — University of the Basque Country (UPV/EHU); Elena Ruiz de Gopegui Palacios, Principal Investigator — University of the Basque Country (UPV/EHU); Miren Vilor Fernandez, Study Chair — University of the Basque Country (UPV/EHU); Ana Garcia de la Fuente, Study Chair — University of the Basque Country (UPV/EHU); Ruth Estefania Fresco, Study Chair — University of the Basque Country (UPV/EHU); Xavier Marichalar Mendia, Study Chair — University of the Basque Country (UPV/EHU)
Locations (1):
- Department fo Stomatology II, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study will be identified by a code and only the researcher will be able to relate them. The personal data will be treated with absolute confidentiality in accordance with the Data Protection Law and will remain in the patient's clinical history. The coded data will be included in a UPV/EHU´s file with reference number 2080310015-INA0110, whose head is Ana María García de la Fuente, and will only be used for the purposes of this project.

REFERENCES:
- [Background] Buti J, Baccini M, Nieri M, La Marca M, Pini-Prato GP. Bayesian network meta-analysis of root coverage procedures: ranking efficacy and identification of best treatment. J Clin Periodontol. 2013 Apr;40(4):372-86. doi: 10.1111/jcpe.12028. Epub 2013 Jan 24. PMID 23346965
- [Background] Cairo F, Nieri M, Cincinelli S, Mervelt J, Pagliaro U. The interproximal clinical attachment level to classify gingival recessions and predict root coverage outcomes: an explorative and reliability study. J Clin Periodontol. 2011 Jul;38(7):661-6. doi: 10.1111/j.1600-051X.2011.01732.x. Epub 2011 Apr 20. PMID 21507033
- [Background] Cairo F, Pagliaro U, Nieri M. Treatment of gingival recession with coronally advanced flap procedures: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):136-62. doi: 10.1111/j.1600-051X.2008.01267.x. PMID 18724847
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Griffin TJ, Cheung WS, Zavras AI, Damoulis PD. Postoperative complications following gingival augmentation procedures. J Periodontol. 2006 Dec;77(12):2070-9. doi: 10.1902/jop.2006.050296. PMID 17209793
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424
- [Background] Esteibar JR, Zorzano LA, Cundin EE, Blanco JD, Medina JR. Complete root coverage of Miller Class III recessions. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):e1-7. PMID 21837295
- [Background] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743
- [Background] Sanz M, Lorenzo R, Aranda JJ, Martin C, Orsini M. Clinical evaluation of a new collagen matrix (Mucograft prototype) to enhance the width of keratinized tissue in patients with fixed prosthetic restorations: a randomized prospective clinical trial. J Clin Periodontol. 2009 Oct;36(10):868-76. doi: 10.1111/j.1600-051X.2009.01460.x. Epub 2009 Aug 12. PMID 19678861
- [Background] Nevins M, Nevins ML, Kim SW, Schupbach P, Kim DM. The use of mucograft collagen matrix to augment the zone of keratinized tissue around teeth: a pilot study. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):367-73. PMID 21837302
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Result] McGuire MK, Scheyer ET. Long-Term Results Comparing Xenogeneic Collagen Matrix and Autogenous Connective Tissue Grafts With Coronally Advanced Flaps for Treatment of Dehiscence-Type Recession Defects. J Periodontol. 2016 Mar;87(3):221-7. doi: 10.1902/jop.2015.150386. Epub 2015 Oct 15. PMID 26469812
- [Result] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988
- [Result] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Result] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Result] Molnar B, Aroca S, Keglevich T, Gera I, Windisch P, Stavropoulos A, Sculean A. Treatment of multiple adjacent Miller Class I and II gingival recessions with collagen matrix and the modified coronally advanced tunnel technique. Quintessence Int. 2013 Jan;44(1):17-24. doi: 10.3290/j.qi.a28739. PMID 23444157
- [Result] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Coronally advanced flap with and without a xenogenic collagen matrix in the treatment of multiple recessions: a randomized controlled clinical study. Int J Periodontics Restorative Dent. 2014;34 Suppl 3:s97-102. doi: 10.11607/prd.1605. PMID 24956099
- [Result] Atieh MA, Alsabeeha N, Tawse-Smith A, Payne AG. Xenogeneic collagen matrix for periodontal plastic surgery procedures: a systematic review and meta-analysis. J Periodontal Res. 2016 Aug;51(4):438-52. doi: 10.1111/jre.12333. Epub 2015 Nov 7. PMID 26547393
- [Derived] Elena RD, Miren VF, Ana-Maria GD, Xabier MM, Luis-Antonio AZ. Analysis of the treatment of RT2 recessions with a xenogeneic collagen matrix vs. connective tissue graft combined with a coronally advanced flap. A double-blinded randomized clinical trial. Clin Oral Investig. 2024 Mar 15;28(4):215. doi: 10.1007/s00784-024-05602-9. PMID 38489063